CLINICAL TRIAL: NCT05001334
Title: Evaluating the Efficiency of Kangaroo Care on Physiological Weight Loss in Term Newborns by Means of Number of Feedings, Number of Diapers and Periodic Weight Measurements
Brief Title: Effect of Kangaroo Care on Phyiological Weight Loss in Term Newborns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Nuray Dilek, Nurse, MSc, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Kanguru
Record Dates: First submitted 2021-06-09; First posted 2021-08-11 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Infant, Newborn; Weight Loss
Keywords: term newborn; weight loss; kangaroo care
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kangaroo care (Experimental): The mothers of the experimental group who accept to participate in the research are given training on how to make kangaroo care and what to pay attention to.
  Interventions: Behavioral: Kangaroo care training
- Control group (No Intervention): The mothers of the control group who accept to participate in the research are NOT given any extra training other than routine breastfeeding and care of a newborn.

INTERVENTIONS:
Behavioral: Kangaroo care training — During perinatal period, mothers are given extra training (other than routine newborn care) about kangaroo care. Baby-mother diad is called for weight check-ups.
  Arms: Kangaroo care

SUMMARY:
The aim of the study is to evaluate the effect of kangaroo care on physiological weight loss in term newborns.

DETAILED DESCRIPTION:
The data collection process continues in a randomized controlled experimental study conducted to determine the effect of kangaroo care on physiological weight loss in term newborns. In the calculation made for the determined effect size, 80% power, 5% margin of error and one-way statistical significance, the experimental group was planned as 51 and the control group as 51 newborns. In this reporting period, 25 newborns as the experimental group and 30 newborns as the control group were followed up and interviewed with the mother.

Mothers who meet the criteria to participate in the research are informed about the research in the delivery room or in the first hours of delivery. The mothers of the experimental group who accept to participate in the research are given training on how to make kangaroo care and what to pay attention to.

Breastfeeding of the mother, the number and frequency of bottle feeding, kangaroo care, diuresis, defecation numbers and weight are recorded by following up. Physiological weight losses are determined by comparing birth weight with daily weight losses.

A cotton kangaroo care blanket is given to every mother who agrees to participate in the study, so that mothers can care for their kangaroos comfortably and to continue kangaroo care at home. These covers, prepared for kangaroo care, increase the motivation of mothers to participate in the study. In order to facilitate the follow-up of diuresis and defecation numbers, the family is supported in the evaluation of diapers (number, weight).

ELIGIBILITY:
Inclusion Criteria:

* Term babies born between 37-42 weeks of gestation
* Newborns born vaginally
* Newborns with developed sucking and swallowing reflexes

Exclusion Criteria:

* Newborns born with C-section
* Newborns in need of NICU care
* Preterm newborns (born <37 weeks of gestation)
* Newborns in need of oxygen
* Genetic or metabolic disease (of the baby) limiting breastfeeding
* HIV (+) mother
* Mother having a chronic disease that will affect breastfeeding
* Mother using drugs that pass into the breastmilk and affect the baby
* Presence of a medical problem that will prevent the mother and baby from staying together

Max Age: 1 Week | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 102 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Physiological weight loss evaluation | 1 week
  Physiological weight loss of term newborns whose mothers are trained about and perform kangaroo care, is theorised to be less than those who receive standard newborn care information. Periodical weight measurements will be recorded. To evaluate feeding efficiency, number of feedings and kangaroo care periods, changed diaper numbers will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa Florence Nightingale School of Nursing, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
If required participant information can be shared